CLINICAL TRIAL: NCT06788340
Title: MOdel-Informed Precision Dosing (MIPD) of Ustekinumab and VEdolizumab in Inflammatory Bowel Disease - An Independent Randomized Controlled Trial
Brief Title: MOdel-Informed Precision Dosing of Ustekinumab and VEdolizumab in Inflammatory Bowel Disease
Acronym: MOVE-IT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32844; 2024-517123-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-07; First posted 2025-01-23 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: MIPD; Model-Informed Precision Dosing; Therapeutic Drug Monitoring; TDM; Inflammatory Bowel Disease; Crohn's disease; Ulcerative colitis; Biologic therapy; Ustekinumab; Vedolizumab
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Model-informed precision dosing of Vedolizumab/Ustekinumab (Experimental): Patients will have blood- and stool samples collected, as well as date and time of drug administration every 4th week. All of these informations, in addition to some informations collected at inclusion, will be used in a PK-model to prescribe when the next dosage of drug should be administered to keep the patient in the therapeutic window.
  Interventions: Drug: PK-model to decide when to dose Vedolizumab and Ustekinumab
- Dosing of Vedolizumab/Ustekinumab by physicians best clinical assessment (No Intervention): Patients will have blood- and stool samples collected every 4 weeks, but these will be blinded for the physicians. They are to be treated as regular patients, but will be seen every 24 weeks to collect clinical activity scores, register alterations in concomitant medication and possible serious adverse events.

INTERVENTIONS:
Drug: PK-model to decide when to dose Vedolizumab and Ustekinumab — the pharmacokinetic model will include information about inflammatory parameters both in blood- and fecal samples, as well as weight, sex, previous treatments and drug concentration.
  Arms: Model-informed precision dosing of Vedolizumab/Ustekinumab

SUMMARY:
The goal of this clinical trial is to investigate if dosage of Ustekinumab (UST) and Vedolizumab (VDZ) based on Model-Informed Precision Dosing (MIPD) is equally as efficient in keeping adults with Inflammatory Bowel Disease (IBD) in remission as management based on what the treating physician deems best. The main question is:

Is using pharmacokinetic-pharmacodynamic (PK-PD) models to predict the appropriate dose and dosing interval for VDZ and UST at least as effective as current practices in maintaining IBD remission.

As above mentioned the comparison-group is adults with IBD, treated with UST or VDZ, managed as the physician deems best.

Participants will:

Have blood and stool tests done, as well as answer a questionnaire 4th weekly Have their dosage frequency decided on either by the PK-model or as the physician deems best visit the clinic once every 24 weeks for checkups. Have an endoscopy done at completion of the study (if the disease is primarily located in the small intestine, MRI or capsule endoscopy will be used instead)

DETAILED DESCRIPTION:
Patients will 4th weekly have their drug-concentration in blood measured (and if low, also antidrug antibodies). Hemoglobin, Albumin, CRP and white blood cell count will also be done, as well as a stool-sample for calprotectin measurement.

For the control group however, the clinicians and patients will be blinded for the results of the blood- and stool samples, and the samples for drug concentration will not get analyzed before end of study.

4th weekly they will also answer PRO2 questionnaire, as well as the VAS-F. 8th weekly they will in addition to above mentioned also answer the EQ-5D-5L questionnaire.

At inclusion, after 24 weeks, and at 48 weeks the patients will in addition to the above mentioned also answer the short IBDQ and WPAI questionnaires, as well as be seen in the outpatient clinic to obtain HBI or SCCAI score as applicable, as well as to document any changes in concomitant medication or diseases, and to register if any serious adverse events have presented.

At completion of the trial, patients will have a endoscopy done.

In one subprotocol, the investigators will include 20 patients from Odense to have an endoscopy at both inclusion and completion. Here they will also have biopsies taken from all segments of the colon, which will be stores in a biobank for future research.

In another subprotocol 20 patients will be included to have a intestinal ultrasound done at inclusion and completion.

In a biobank for future research the investigators will also store serum-samples, buffy coat, and stool samples collected at inclusion, after 24 and 48 weeks from all included patients.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis or Crohn's disease. Diagnosed, according to universally acknowledged criteria, a minimum of 3 months prior to inclusion
* Age ≥ 18
* Stable treatment with VDZ or UST for at least 3 months prior to inclusion
* Stable disease activity, mild activity is accepted, defined by fecal calprotectin ≤ 200, and a weighted PRO2 < 14 for CD or a PRO2 ≤3 for UC
* No change in medical therapy within 3 months prior to inclusion, as concomitant therapy with other immune suppressants is allowed (Azathioprine, 6-mercaptopurine, Methotrexate, 5-aminosalicylic acid)
* The patient must be able to understand patient information material
* The patient must be able to give informed written consent

Exclusion Criteria:

* Having a diagnose of indeterminate colitis
* Having a stoma or pouch
* Fistulizing disease being the primary reason for treatment with VDZ or UST
* Expected eminent change of therapy
* Expected need for surgical intervention within the coming 3 months
* Contraindication against continuing treatment with VDZ or UST, including prior acute or delayed infusion reaction to VDZ or UST
* Any active infection requiring parenteral treatment, known infection with tuberculosis, human immunodeficiency virus (HIV) or hepatitis virus.
* Any condition which the responsible physician finds incompatible with participation in the study
* Patients unable to participate in the collection of symptoms scores
* Patients who are pregnant or nursing at time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
The fraction of patients in steroid-free remission | at the end of the observation period (48 weeks)
  ((for CD defined by PRO2 ≤ 4, for UC defined by PRO2 = 0) AND a fecal calprotectin ≤200)

SECONDARY OUTCOMES:
The fraction of the observation period (48 weeks) where the disease is in steroid-free remission | this is registered every 4th week throughout the study duration of 48 weeks.
  for CD defined by patient reported outcome 2 (PRO2) stool frequency <= 3 and abdominal pain < = 1, for UC defined by PRO2, number of abnormal stools for the patient, bleeding from the rectum = 0) AND a fecal calprotectin ≤ 200.
The financial costs associated with the two treatment strategies over the observation period (12 months) | through study completion, an average of 48 weeks
  expenditure on medicines (both expenditure on the purchase of medicines and expenditure on the administration of medicines), expenses for doctor visits / visits to a nurse, possibly expenses for hospitalization, possibly expenses for surgery, possibly expenses for sick leave and possibly expenses for early retirement.
  After end of study, the investigators will collect data on sick leave etc. from the national patient registry.
Endoscopic healing of the mucosa | at completion of study, approximately 48 weeks
  for CD assessed by Simple Endoscopic Score for Crohn's Disease (SES-CD) <3; and for UC assessed on the basis of the Ulcerative Colitis Endoscopic Index of Severity (UCEIS)≤1. If disease is primarily located in the small intestine, MRI or capsule endoscopy will be used instead, and assessed by the simplified MaRIA score <1 or Lewis score ≤135, respectively
Changes in quality of life during the study period | 48 weeks
  assessed by Short Inflammatory Bowel Disease Questionnaire (SIBDQ) difference between baseline and end of study. Improvement of quality of life indicated by a positive change of the SIBDQ. SIBDQ is collected at inclusion, week 24 and week 48. A higher the score, indicates a better outcome, Maksimum score of 70 points.
Quality of life as QALYs | 48 weeks
  assessed by the EuroQol-5 dimensions-5 levels questionnaire (EQ-5D-5L) and converted to QALYs. The cost per QALY will also be calculated. EQ-5D-5L is collected every 8th week throughout the study. Score ranges from 5-25, a higher score indicating poorer quality of life.
Clinical Disease Activity | 48 weeks
  assessed by Simplified Clinical Colitis Activity Index (SCCAI) for UC and Harvey-Bradshaw Index (HBI) for CD. These are collected at inclusion and every 24th week thereafter. SCCAI score ranges from 0-19, a higher score indicating a more severe disease activity. HBI score ranges from 0-20, a higher score indicating more severe disease activity.
Inflammatory burden over the observational period | 48 weeks
  CRP, albumin, hemoglobin, leukocyte counts and fecal calprotectin. These will be collected every 4th week
Expenses for analysis of drug concentration | 48 weeks
  patients will have drug concentrations analyzed every 4th week, the price of this will be collected
Expenses for drugs | 48 weeks
  patients will typically administer sc VDZ every 4th to 2nd week, iv VDZ every 12th to 4th week and UST every 12th to 4th week
Drug persistency | 48 weeks
  number of patients switching to another treatment during the study
Disease flares | 48 weeks
  assessed by consumption of glucocorticoids or IBD-related surgery
Fatigue | 48 weeks.
  to assess if treating according to a PK-model results in less fatigue measured by Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F). Patients are asked to register how fatigued they feel every 4th week throughout the study. The VAS-F is a visual analogue scale that goes from 0-10, 10 indicating severe fatigue.
Disease impact on work productivity and performance of daily activities | 48 weeks
  Assessed by difference in Work Productivity and Activity Impairment questionnaire (WPAI) scores and changes in scores between patients in the intervention- and control group. WPAI is collected at inclusion and every 24th week throughout the study.
  WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Ainsworth, professor, DMSc, Principal Investigator — Odense University Hospital
Locations (6):
- Denmark (6):
  - Dept. of Gastrointestinal Diseases, Aalborg
  - Dept. of Internal Medicin, Esbjerg
  - Dept. of Gastrointestinal Diseases, Hvidovre
  - Dept. of medicine, Nyborg
  - Dept. of Gastrointestinal Diseases, Odense
  - Dept. of Medicine, Vejle

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will possibly be shared, including clinical characteristics, laboratory test results, and patient-reported outcomes relevant to the study endpoints.
  Data will be available after publication of the main trial results and completion of any relevant follow-up studies. This is expected to occur approximately one year after the study's primary completion date.
  Data will be available for a minimum of 5 years following the publication of the trial results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: will become available approximately March 2028 and will be available for at least 5 years
Access Criteria: Data will be shared with qualified researchers conducting legitimate scientific inquiries, particularly those working within the field of inflammatory bowel disease (IBD) and therapeutic drug monitoring (TDM)

REFERENCES:
- [Derived] Frimor C, Steenholdt C, Widigson ESK, Kjeldsen J, Larsen L, Burisch J, Joergensen MT, Halling ML, Kloft C, Ainsworth MA. MOdel-informed precision dosing (MIPD) of ustekinumab and VEdolizumab in inflammatory bowel disease: protocol for an Independent randomised, controlled, multicentre Trial (MOVE-IT). BMJ Open Gastroenterol. 2025 Dec 25;12(1):e001985. doi: 10.1136/bmjgast-2025-001985. PMID 41453773